CLINICAL TRIAL: NCT05399225
Title: Comparison Between Platelets to Lymphocytes Ratio and Procalcitonin in Prediction of Sepsis Outcome
Brief Title: Platelets to Lymphocytes Ratio in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Elmalah, assistant lecturer, Tanta University
Other Study IDs: Platelets to lymphocytes ratio
Record Dates: First submitted 2021-08-28; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Platelets to Lymphocytes Ratio Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platelets to lymphocytes ratio and procalcitonin: Platelets to lymphocytes ratio in patients with sepsis
  Interventions: Diagnostic Test: Platelets to lymphocytes ratio and procalcitonin
- Procalcitonin group: Procalcitonin in patient with sepsis
  Interventions: Diagnostic Test: Platelets to lymphocytes ratio and procalcitonin

INTERVENTIONS:
Diagnostic Test: Platelets to lymphocytes ratio and procalcitonin — Platelets to lymphocytes ratio and procalcitonin in sepsis

SUMMARY:
The aim of this study is to compare effectiveness of platelets to lymphocytes ratio (PLR) with procalcitonin as a predictor of sepsis outcome.

DETAILED DESCRIPTION:
Sepsis is a rapidly progressive, life-threatening disease. Accurate and expeditious assessment of sepsis is important for early administration of antibiotics and removal of the source of infection.

In the 2016 version of the sepsis guidelines (Sepsis-3), the concept of the systemic inflammatory response syndrome has been deleted.

Although most patients with sepsis receive intensive management, such as early goal directed therapy (EGDT), in an emergency department (ED), the mortality rate of sepsis has been reported to be greater than 20% to 30%.

Many clinicians have studied the usefulness of blood biomarkers such as C-reactive protein, procalcitonin, and lactate for early assessment of sepsis and for prognostication, in order to initiate timeous treatment and to prevent rapid progression to multi-organ failure.

Several studies mentioned the advantages of the precursor molecule of calcitonin, namely procalcitonin as a biomarker for sepsis.

In recent years, studies have reported that platelets and lymphocytes play critical roles in the inflammatory process. Therefore, the platelet-to-lymphocyte ratio (PLR) a novel inflammatory factor has received research attention recently, as it may act as an indicator of inflammation, in a wide spectrum of diseases, such as myocardial infarction,acute kidney injury (AKI), Based on the findings of previous studies, it is reasonable to speculate the presence of a potential relationship between PLR and mortality for sepsis.

Platelet to lymphocytes ratio is defined as the ratio of the absolute platelet count and absolute lymphocyte count.

ELIGIBILITY:
Inclusion Criteria:

1. Septic patients according to Third International Consensus Definitions for Sepsis
2. with ICU stay more than 24 hours will be included.

Exclusion Criteria:

1. Pregnant and women in puerperium.
2. Patients with active hemorrhage
3. Patients with hematological diseases (including bone marrow diseases) and collagen diseases.
4. Patients on corticosteroid therapy or immunosuppressive drugs.
5. Patients who will need immediate surgical interventions.
6. Acute cerebrovascular or coronary syndrome.
7. Patients received blood or platelets transfusion before enrollment in the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross sectional
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The prediction of 28 days mortality. | during 28 days from patient admission till patient discharge or death.
  Prediction of 28 days mortality in icu patients with sepsis according to change in platlet to lymphocyte ratio

SECONDARY OUTCOMES:
Length of icu stay | throught study comletion, maximum 28 days
  number of days that past during patient presence in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university of medicine, Tanta, Egypt